CLINICAL TRIAL: NCT02267772
Title: A Randomized, Controlled Trial of IV Acetaminophen Versus IV Morphine to Manage Pain in Pregnancy: Can Opioid Use be Reduced in Pregnant Women?
Brief Title: IV Acetaminophen vs IV Morphine for Pain Control in Pregnant Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruitment
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jerrie Refuerzo, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-13-0763
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Pain Management in Pregnant Women
MeSH Terms: interventions — Acetaminophen; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Acetaminophen (Experimental): IV acetaminophen for pain control
  Interventions: Drug: IV Acetaminophen
- IV morphine (Active Comparator): IV morphine for pain control
  Interventions: Drug: IV Morphine

INTERVENTIONS:
Drug: IV Acetaminophen — IV Acetaminophen
  Arms: IV Acetaminophen
Drug: IV Morphine — IV Morphine
  Arms: IV morphine

SUMMARY:
Purpose: To determine if IV acetaminophen can 1) decrease pain in pregnancy women, 2)reduce the amount of opioid use in pregnant women who encounter pain, 3) reduce maternal and fetal adverse effects compared to opioids.

Design: This is a comparative effective trial that is a randomized, controlled trial of IV acetaminophen vs. IV morphine in pregnant women.

Procedures: Women meeting inclusion/exclusion criteria will be randomized to IV acetaminophen or IV morphine. The IV acetaminophen group will get up to four standard doses of IV acetaminophen during their stay at the hospital. The second group will get up to six standard doses of morphine. Subjects will complete a pain scale after medication administration and will be asked about any side effects.

DETAILED DESCRIPTION:
Rationale for this clinical trial The goal of analgesia in pregnancy is to reduce pain while minimizing both maternal and fetal adverse effects. Current opioids used in pregnancy provide minimal pain relief and are associated with adverse effects. IV acetaminophen has been shown to significantly improve pain control following cesarean section and in the first stage of labor. Moreover, IV acetaminophen reduces the need and consumption of opioids following surgery. If IV acetaminophen can be as effective in controlling pain associated with maternal medical conditions and uterine contractions with labor, then the use of parenteral opioids in pregnant women and its exposure to the fetus could be reduced. This could provide new opportunities in the medical management of pain in pregnancy. Thus we propose a comparative effectiveness trial of IV acetaminophen compared to IV morphine.

Hypothesis:

We hypothesize that IV acetaminophen is as effective as IV morphine in reducing pain in pregnant women. In doing so, IV acetaminophen can reduce the amount of narcotics needed in women with pain.

Objectives:

To determine if IV acetaminophen can:

1. Decrease pain in pregnant women
2. Reduce the amount of opioid use in pregnant women who encounter pain
3. Reduce maternal and fetal adverse effects compared to opioids

Study Design:

For this comparative effective trial, we propose a randomized, controlled trial of IV acetaminophen vs. IV morphine in pregnant women. Prior studies have confirmed that IV acetaminophen is effective in controlling pain compared to placebo.[14,20] Thus, administering just a placebo for pain control is not justified at this time.

We will include 3 different groups of pregnant populations who encounter pain for different reasons.

Group 1: Pregnant women with uterine contractions, but not in labor Group 2: Pregnant women with uterine contractions in the first stage of labor Group 3: Pregnant women with a medical condition associated with pain.

ELIGIBILITY:
Inclusion criteria:

Group 1. We will include pregnant women greater than 24 weeks of pregnancy who present with uterine contractions, but are not in labor and who are warranting treatment with intravenous medication for pain control as part of their routine treatment. This will be defined as the presence of uterine contractions documented on the tocodynamometer. However, the cervix remains less than 2 cm dilated and has not changed after 1 hour after re-examining her cervix.[23]

Group 2. We will include pregnant women greater than 34 weeks of pregnancy who present with uterine contractions and are in the first stage of labor and who are warranting treatment with intravenous medication for pain control as part of their routine treatment. This will be defined as the presence of uterine contractions documented on the tocodynamometer and cervical dilation greater than 2 cm, but less than 6 cm. [23]

Group 3. We will include pregnant women greater than 16 weeks of pregnancy who present with pain due to a maternal medical condition including sickle cell crisis, pyelonephritis, pancreatitis, cholecystitis, nephrolithiasis or headache and who are warranting treatment with intravenous medication for pain control as part of their routine treatment.

Exclusion criteria:

We will exclude women less than 18 years of age, less than 16 weeks gestation, with weight less than 50 kg, and contraindications to acetaminophen including reported elevated liver function tests, hepatic injury, hepatic disorder, active liver disease, alcoholism, chronic malnutrition, known coagulopathy, hemorrhage, creatinine > 1.0, or known allergy or hypersensitivity to acetaminophen. We will also exclude women who have received any opioids within the last 24 hours.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2014-01; Primary Completion 2019-04-27 (Actual); Study Completion 2019-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerrie S Refuerzo, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Lyndon B Johnson Hospital, Houston, Texas
  - Memorial Hermann Hospital, Texas Medical Center, Houston, Texas

REFERENCES:
- [Derived] Ankumah NE, Tsao M, Hutchinson M, Pedroza C, Mehta J, Sibai BM, Chauhan SP, Blackwell SC, Refuerzo JS. Intravenous Acetaminophen versus Morphine for Analgesia in Labor: A Randomized Trial. Am J Perinatol. 2017 Jan;34(1):38-43. doi: 10.1055/s-0036-1584143. Epub 2016 May 16. PMID 27182992

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 163 were enrolled, including those in Group 1 (Pregnant women with uterine contractions, but not in labor), Group 2 (Pregnant women with uterine contractions in the first stage of labor), and Group 3 (Pregnant women with a medical condition associated with pain). The participant flow only reflects participants enrolled in Group 1 and Group 2, and not those in Group 3.
Period: Overall Study
Arm/Group | IV Acetaminophen | IV Morphine
Started | 50 | 52
Randomized | 50 | 52
Received Study Drug | 48 | 52
Completed | 48 | 52
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Acetaminophen | IV Morphine | Total
Number analyzed (Participants) | 48 | 52 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.0 (5.5) | 27.5 (6.0) | 27.3 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 100
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black | 19 | 24 | 43
  Caucasian | 5 | 8 | 13
  Hispanic | 19 | 21 | 40
  Other | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 48 | 52 | 100

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Intensity as Assessed by a Visual Analogue Scale (VAS)
Description: The visual analogue scale (VAS) ranges from 0mm to 140mm. The subject will be asked to mark with a pen on the scale to rate their pain. Negative differences in scores indicated a pain score worse than baseline and positive differences indicated an improved pain score from baseline.
Time Frame: baseline, 120 minutes after administration
Population: For the IV Acetaminophen arm, data were collected for 24 out of 30 participants in pre-labor and 18 out of 18 participants in the 1st stage of labor. For the IV morphine arm, data were collected for 30 out of 32 participants in pre-labor and 20 out of 20 participants in the 1st stage of labor.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IV Acetaminophen | IV Morphine
Number analyzed (Participants) | 42 | 50
score on a scale
  pre-labor group: number analyzed (Participants) | 24 | 30
  pre-labor group | 2.67 (3.8) | 3.2 (5.1)
  first stage of labor group: number analyzed (Participants) | 18 | 20
  first stage of labor group | -18.2 (13.2) | -4.8 (12.5)

2. Secondary Outcome: Pain Relief Based on a 5 Point Verbal Scale
Time Frame: 24 hrs
Population: Data were not collected for this outcome measure.
Arm/Group | IV Acetaminophen | IV Morphine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants Who Received Rescue Medications
Time Frame: 24 hours after administration
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | IV Morphine
Number analyzed (Participants) | 50 | 52
Participants | 30 | 19

4. Secondary Outcome: Quantity of Rescue Medication Over 24 Hours
Time Frame: 24 hours after administration
Population: Data were not collected for this outcome measure.
Arm/Group | IV Acetaminophen | IV Morphine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Total Amount of Study Drug Administered
Time Frame: 24 hours after administration
Population: For the IV Acetaminophen arm, data were collected for 30 out of 30 participants in pre-labor and 18 out of 18 participants in the 1st stage of labor. For the IV morphine arm, data were collected for 32 out of 32 participants in pre-labor and 20 out of 20 participants in the 1st stage of labor.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | IV Acetaminophen | IV Morphine
Number analyzed (Participants) | 48 | 52
milligrams
  pre-labor group: number analyzed (Participants) | 30 | 32
  pre-labor group | 1600 (952.2) | 6.4 (1.9)
  1st stage of labor group: number analyzed (Participants) | 18 | 20
  1st stage of labor group | 1055 (229) | 2.3 (0.72)

6. Secondary Outcome: Patient's Global Satisfaction at 24 Hours
Description: This will be patient reported.
Time Frame: 24hrs
Population: Data were not collected for this outcome measure.
Arm/Group | IV Acetaminophen | IV Morphine
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Maternal Side Effects
Description: Maternal side effects include nausea, vomiting, headache, pruritus, insomnia, and drowsiness.
Time Frame: 1 hour after administration
Population: Data for this outcome measure were not collected for 5 in the IV Acetaminophen arm and 1 in the IV morphine arm.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | IV Morphine
Number analyzed (Participants) | 43 | 51
Participants
  nausea | 2 | 2
  vomiting | 0 | 3
  headache | 5 | 6
  pruritus | 2 | 4
  insomnia | 5 | 7
  drowsiness | 17 | 15

8. Secondary Outcome: Number of Participants With Fetal Heart Rate Changes
Description: Changes in fetal heart rate tracing include acceleration, decelerations, and variability.
Time Frame: 1 hour after administration
Population: Data for this outcome measure were not collected for 6 in the IV Acetaminophen arm and 4 in the IV morphine arm.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Acetaminophen | IV Morphine
Number analyzed (Participants) | 42 | 48
Participants
  absence of accelerations | 4 | 12
  late decelerations | 1 | 1
  minimal or absent variability | 4 | 3

ADVERSE EVENTS:
Time Frame: 1 hour after administration
Description: Other (Not Including Serious) Adverse Events were not collected for 5 in the IV Acetaminophen arm and 1 in the IV morphine arm. All participants who study drug were assessed for serious adverse events (SAEs) and Mortality.
Arm/Group | IV Acetaminophen | IV Morphine
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/48 | 0/52
Other Adverse Events (participants affected / at risk) | 21/43 | 15/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Acetaminophen (N=48) | IV Morphine (N=52)
Adverse reaction to demerol administered as rescue medication, which required narcan for reversal (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Acetaminophen (N=43) | IV Morphine (N=51)
Nausea (General disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Headache (General disorders) | 5 (5) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Insomnia (General disorders) | 5 (5) | 7 (7)
Drowsiness (General disorders) | 17 (17) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT02267772/Prot_SAP_000.pdf